CLINICAL TRIAL: NCT06659640
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled, 2-part Study of the Safety, Tolerability, Efficacy, Pharmacokinetics, and Pharmacodynamics of Single Dose ALN-6400 in Adult Healthy Volunteers and Multiple Dose ALN-6400 in Adult Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: A Study to Evaluate ALN-6400 in Healthy Volunteers and Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-6400-001; 2025-522510-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: siRNA; RNAi therapeutic; Plasminogen; PLG; HHT; Osler-Weber-Rendu; epistaxis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: ALN-6400 (Experimental): Participants will be administered a single dose of ALN-6400.
  Interventions: Drug: ALN-6400
- Part A: Placebo (Placebo Comparator): Participants will be administered a single dose of placebo.
  Interventions: Drug: Placebo
- Part B: ALN-6400 (Experimental): Participants will be administered multiple doses of ALN-6400.
  Interventions: Drug: ALN-6400
- Part B: Placebo (Placebo Comparator): Participants will be administered multiple doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-6400 — ALN-6400 will be administered subcutaneously (SC)
  Arms: Part A: ALN-6400; Part B: ALN-6400
Drug: Placebo — Placebo will be administered subcutaneously (SC)
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to:

* evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending doses of ALN-6400 in healthy volunteers
* evaluate the efficacy, safety, tolerability and PD of multiple doses of ALN-6400 in adult patients with HHT

ELIGIBILITY:
Inclusion Criteria -

Part A:

* Is a healthy adult volunteer

Part B:

* Is an adult patient with a clinical diagnosis of HHT

Exclusion Criteria -

Part A:

* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN)
* Has known human immunodeficiency virus (HIV) infection; or known current or chronic hepatitis C virus or hepatitis B virus infection
* Has an estimated glomerular filtration (eGFR) of <90 mL/min/1.73m^2 at screening

Part B:

* Has ALT or AST >2×ULN
* Has total bilirubin >1.5×ULN
* Has eGFR of <30 mL/min/1.73m^2 at screening

Parts A and B:

* Is not willing to comply with the contraceptive requirements during the study period

Note: other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2028-01-05 (Estimated); Study Completion 2028-06-22 (Estimated)

PRIMARY OUTCOMES:
Part A: Frequency of Adverse Events | Up to Week 36
Part B: Frequency of Adverse Events | Up to Week 96

SECONDARY OUTCOMES:
Part A: Concentrations of ALN-6400 in Plasma | Predose and up to 2 days postdose
Part A: Change from Baseline in Plasminogen (PLG) in Plasma Protein Levels | Predose and up to Week 36 postdose
Part B: Change from Baseline in Plasminogen (PLG) in Plasma Protein Levels | Screening and up to Week 96 postdose
Part A: Change from Baseline in Plasminogen (PLG) in Plasma Activity Levels | Predose and up to Week 36 postdose
Part B: Change from Baseline in Plasminogen (PLG) in Plasma Activity Levels | Part B: Screening and up to Week 96 postdose
Part B: Change from Baseline in Intensity-adjusted Epistaxis Duration | Baseline up to Week 96
  Intensity-adjusted epistaxis duration will be assessed using a daily patient epistaxis diary.
Part B: Change from Baseline in Epistaxis Severity Score (ESS) Scale | Baseline up to Week 96
  Validated bleeding scale in HHT scored between 0-10, higher scores indicate worse bleeding.
Part B: Change from Baseline in Epistaxis Duration | Baseline up to Week 96
  Epistaxis duration will be assessed using a daily patient epistaxis diary.
Part B: Change from Baseline in Epistaxis Frequency | Baseline up to Week 96
  Epistaxis frequency will be assessed using a daily patient epistaxis diary.
Part B: Change from Baseline in Epistaxis Intensity | Baseline up to Week 96
  Epistaxis intensity will be assessed using a daily patient epistaxis diary.
Part B: Change from Baseline in Epistaxis-free Days per Month | Baseline up to Week 96
  Epistaxis-free days per month will be assessed using a daily patient epistaxis diary.
Part B: Change from Baseline in Hematologic Support Score (HSS) | Baseline up to Week 96
  The HSS is a quantitative tool designed to longitudinally assess the red blood cells (RBC) and iron supplementation needs of patients with HHT and other chronic bleeding disorders.
Part B: Change from Baseline in Iron Infusions | Baseline up to Week 96
Part B: Change from Baseline in Red Blood Cell (RBC) Infusions | Baseline up to Week 96
Part B: Change from Baseline in Hemoglobin | Baseline up to Week 96
Part B: Change from Baseline in Quality of Life Patient-reported Outcomes (QoL/PRO) assessed by Nasal Outcome Score for Epistaxis in Hereditary Hemorrhagic Telangiectasia (NOSE HHT) Score | Baseline up to Week 84
  HHT-specific QoL/PRO will be assessed using the NOSE HHT score. The NOSE HHT is a 29-item patient-reported, clinically validated outcome measure, with total scores ranging continuously from 0 to 4 with higher scores indicating worse scores.
Part B: Change from Baseline in QoL/PRO assessed by Modified Patient Global Impression of Severity (mPGI-S) Score | Baseline up to Week 84
  HHT-specific QoL/PRO will be assessed using the mPGI-S. The patient will respond to a single question, providing their global impression of change in their overall status and epistaxis experience.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (8):
- United States (2):
  - Clinical Trial Site, Cypress, California
  - Clinical Trial Site, Boston, Massachusetts
- Canada (2):
  - Clinical Trial Site, Mount Royal
  - Clinical Trial Site, Toronto
- France (2):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Bron
- Clinical Trial Site, Homburg, Germany
- Clinical Trial Site, L'Hospitalet de Llobregat, Spain

IPD SHARING:
Plan to Share IPD: Yes
Phase 2-4:
  Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the United States (US) and/or the European Union (EU).
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.